CLINICAL TRIAL: NCT05845424
Title: Comparison of Efficacy and Safety of High-Intensity Statin and Ezetimibe Combination Versus StanDard carE in AsymptomatiC PatIentS wIth Presence of COroNary Artery CALCIUM (DECISION-CAL)
Brief Title: High-intensity Statin and Ezetimibe Therapy for Asymptomatic Patients With Positive Coronary Calcium
Acronym: DECISION-CAL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seung-Hyuk Choi, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DECISION-CALCIUM
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Calcification; Metabolic Syndrome; Dyslipidemias
MeSH Terms: conditions — Metabolic Syndrome; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: standard treatment vs. aggressive treatment
Masking Description: A prospective, open label, multicenter randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aggressive treatment arm (Experimental): In this group, high-intensity statin (rosuvastatin 20mg) combined with ezetimibe 10 mg will be prescribed regardless of patients' age, concomitant diabetes mellitus, or ASCVD risk.
  Interventions: Drug: High intensity statin plus ezetimibe therapy
- Standard treatment arm (Active Comparator): In this group, lipid lowering therapy will be followed according to the current guideline recommendation. A moderate-intensity statin (rosuvastatin 5 mg) will be prescribed for patients over 75 years of age or with diabetes mellitus. For non-diabetic patients aged 40-75 years, the use of statins will be determined by calculating the ASCVD risk score. (ASCVD risk <7.5%: no statin use, ≥7.5 - <20%: moderate-intensity statin [rosuvastatin 5mg], ≥ 20%: high-intensity statin [rosuvastatin 20mg])
  Interventions: Drug: Guideline directed statin therapy

INTERVENTIONS:
Drug: Guideline directed statin therapy — At least moderate intensity statin, recommended by the current guideline based on the ASCVD risk
  Arms: Standard treatment arm
Drug: High intensity statin plus ezetimibe therapy — Rosuvastatin 20 mg + Ezetimibe 10 mg
  Arms: Aggressive treatment arm

SUMMARY:
The aim of this study is to compare safety and efficacy between the aggressive treatment with combination of high-intensity statin and ezetimibe and the current standard lipid lowering treatment in asymptomatic patients with presence of coronary calcification.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular diseases (ASCVD), such as myocardial infarction (MI), ischemic stroke, or peripheral arterial disease, are the leading cause of morbidity and mortality worldwide. The causality of low-density lipoproteins cholesterol (LDL-C) level in the development of ASCVD is well demonstrated in previous studies. After introducing LDL-C lowering agents, multiple large-scale randomized clinical trials have demonstrated lower cardiovascular events with lowering LDL-C levels. In particular, for secondary prevention, more aggressive control of LDL-C levels with high-intensity statin therapy significantly reduced cardiovascular events compared with moderate-intensity statin therapy. In addition, the Improved Reduction of Outcomes: Vytorin Efficacy International Trial (IMPROVE-IT) proved the clinical efficacy of additive ezetimibe for incrementally lowering of LDL-C levels in patients with acute coronary syndrome. However, there has been limited evidence regarding the efficacy and safety of aggressive lipid-lowering strategy using high-intensity statin with a combination of ezetimibe for primary prevention of cardiovascular events among persons without cardiovascular disease. Although the Heart Outcomes Prevention Evaluation (HOPE)-3 and Justification for the Use of Statins in Prevention: an Intervention Trial Evaluating Rosuvastatin (JUPITER) trials consistently identified that the use of rosuvastatin (10 mg or 20 mg) was significantly associated with reduced future risk of major cardiovascular events in patients who did not have cardiovascular disease, those studies have been focused on the use of statin, not on the intensity of statin.

The coronary artery calcium (CAC) scan, a marker of subclinical coronary atherosclerosis, has become popular for individuals at risk for atherosclerotic cardiovascular disease. CAC is strongly associated with atherosclerotic burden and predicts coronary heart disease events and mortality, regardless of their age, sex, race, or ASCVD risk. Furthermore, the progression of CAC is associated with an increased risk for future hard and total coronary heart disease events. The use of CAC scoring was associated with significant improvements in the reclassification and discrimination of incident ASCVD. Nevertheless, the current guidelines recommend CAC measurement for selected cases only with borderline or intermediate risk of ASCVD to guide the use of statin or not. However, in real-world practice, CAC testing is increasingly being promoted to the public as a means of self-assessment of cardiovascular risk and is widely being used regardless of ASCVD risk. Considering that statin has additional properties, including atherosclerotic plaque stabilization, oxidative stress reduction, enhancement of endothelial function, and a decrease in vascular inflammation beyond their lipid-lowering effect, aggressive treatment with a high-intensity statin plus ezetimibe combination might have beneficial effects on the long-term clinical outcomes for asymptomatic patients with significant coronary calcium (Agatston Score ≥ 100) compared with standard lipid-lowering therapy endorsed by the current guidelines.

Therefore, the purpose of DECISION-CALCIUM (Comparison of Efficacy and Safety of High-Intensity Statin and Ezetimibe Combination versus StanDard carE in AsymptomatiC PatIentS wIth Presence of COroNary Artery CALCIUM) trial is to compare the efficacy and safety of the aggressive lipid-lowering therapy with combination of high-intensity statin and ezetimibe, compared with the current standard lipid-lowering therapy in asymptomatic patients with significant coronary calcification for primary prevention.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 40 years of age.
* Asymptomatic patients with presence of coronary calcification (Agatston Score ≥ 100)
* low-density lipoproteins cholesterol (LDL-C) <190 mg/dL

Exclusion Criteria:

* Objective evidence of at least moderate inducible ischemia requiring revascularization treatment
* History of cerebrovascular disease
* History of coronary or peripheral arterial revascularization
* Active liver disease or persistent unexplained serum transaminase elevations more than 2 times the upper limit of normal range
* History of any adverse drug reaction requiring discontinuation of statin (e, g. rhabdomyolysis)
* Allergy or sensitivity to any statin or ezetimibe
* Concurrent treatment with cyclosporine or a condition likely to result in organ transplantation and the need for cyclosporine
* Pregnancy or breast feeding
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* Unwillingness or inability to comply with the procedures described in this protocol.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  a composite of death from any causes, myocardial infarction, stroke, unplanned coronary revascularization, or other arterial revascularization procedure

SECONDARY OUTCOMES:
All-cause death | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  Death from any causes
Cardiovascular death | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  Death from cardiovascular causes
Stroke | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  Ischemic or hemorrhagic stroke
Unplanned coronary revascularization | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  revascularization procedure to coronary artery
Arterial revascularization procedure | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  All arterial revascularization procedure
Major bleeding | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  Bleeding Academic Research Consortium (BARC) type 3-5
Bleeding | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  BARC type 2-5
Heart failure hospitalization | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  Hospitalization due to heart failure
Coronary calcium progression | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  Delta CAC
Changes of LDL-C | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  Delta LDL-C
New-onset diabetes mellitus | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  Occurence of new-onset diabetes mellitus
Hepatic disorder requiring discontinuation of statin | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  Occurence of hepatic disorder requiring discontinuation of statin
muscle-related adverse events | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  Occurence of muscle-related adverse events due to statin
Proportion of patients with LDL-C < 100mg/dL | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  Proportion of patients with LDL-C < 100mg/dL
Proportion of patients with LDL-C < 70mg/dL | up to 4.5 years of median follow-up (till 3 year after the last patient enrollment)
  Proportion of patients with LDL-C < 70mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hyuk Choi, Principal Investigator — Samsung Medical Center
Locations (1):
- SamsungMedicalCenter, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No